CLINICAL TRIAL: NCT05719207
Title: Efficacy of Balloon Dilation of the Eustachian Tube in Eustachian Tube Dilatory Dysfunction: a Randomized, Sham-controlled Trial
Brief Title: Efficacy of Balloon Dilation of the Eustachian Tube in Eustachian Tube Dilatory Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Justin Lui, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB22-1601
Record Dates: First submitted 2023-01-15; First posted 2023-02-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Eustachian Tube Dysfunction; Barotitis
Keywords: BDET; ETD; ETDD; baro-challenge

STUDY DESIGN:
Intervention Model Description: Parallel design with optional crossover from control to intervention at 6 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Balloon dilation of eustachian tube (Experimental): These patient will undergo balloon dilation dilation of the eustachian tube.
  Interventions: Device: Balloon dilation of eustachian tube
- Sham procedure (Sham Comparator): These patients will undergo a sham procedure, where the motions of balloon dilation of the eustachian tube will be simulated.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Balloon dilation of eustachian tube — Patients in the intervention group would undergo balloon dilation of the eustachian tube under local anesthetic in clinic. The Stryker XprESS LoProfile ENT dilation system or the Stryker Audion ET dilation system will be used.
  Other Names: Stryker XprESS LoProfile ENT dilation system (Stryker ENT, Plymouth, MN, USA.); Stryker Audion ET dilation system (Stryker ENT, Plymouth, MN, USA)
  Arms: Balloon dilation of eustachian tube
Other: Sham procedure — Patients in the sham group will undergo the motions of an in-office dilation of the eustachian tube, without actually dilating the eustachian tube.
  Arms: Sham procedure

SUMMARY:
This study is being conducted to learn more about a procedure, balloon dilation of the eustachian tube, in treating patients with eustachian tube dysfunction. Traditionally, eustachian tube dysfunction is treated with nasal steroid sprays and decongestants, or by placement of ear tubes. However, current evidence suggest that medical options are ineffective, and placement of ear tubes is not risk-free. The investigators are carrying out this research study with the following goals:

1. Determine if balloon dilation of the eustachian tube is superior to a placebo procedure in treating patients with eustachian tube dilatory dysfunction
2. Identify patient variables associated with positive response to balloon dilation of the eustachian tube
3. Re-demonstrate the safety of balloon dilation of the eustachian tube

What does participation in this study involve? Participants in this study will:

* Agree to be randomly assigned to undergo either: balloon dilation of the eustachian tube, or a placebo procedure, with the option to undergo dilation of the eustachian tube 6 weeks later
* Agree to allowing the investigators access to their personal health information
* Complete the following assessments and questionnaires in clinic before undergoing balloon dilation or placebo procedure:

  * A questionnaire to assess your eustachian tube dysfunction
  * An assessment of the movement of your ear drum (tympanogram)
  * A hearing test (audiogram)
  * A questionnaire to assess the impact of eustachian tube dysfunction on work/activity
  * A questionnaire to assess overall health-related quality of life
  * An assessment of the ability to equalize middle ear pressure(s)
  * Visual examination of the ear drums
* Repeat the above assessments and questionnaires over the course of four follow-up appointments at 6-, 24-, and 52-weeks after the procedure.

DETAILED DESCRIPTION:
Adult eustachian tube dilatory dysfunction (ETDD) accounts for over 2 million healthcare visits annually. It can cause longstanding negative middle ear pressure which may lead to otitis media with effusion, tympanic membrane retraction, perforation, middle ear atelectasis and cholesteatoma. Despite this, effective treatments for ETDD are unavailable. Recently, balloon dilation of the eustachian tube (BDET) has gained popularity, where the cartilaginous portion of the Eustachian tube undergoes local dilation with balloon inflation. This technique underwent industry-funded clinical trials in the United States demonstrating its safety and it's superiority to medical management. However, these studies are confounded by industry funding and lack of a blinded control group, the latter of which is critical in a condition where patient-reported outcome measures are relied on. Furthermore, the randomized studies to date do not include patients with baro-challenge ETDD, where symptoms are limited to the context of ambient pressure changes. As such, the investigators opted to perform a non-industry-funded, placebo-controlled trial including both chronic and baro-challenge ETDD patients in a Canadian setting.

Potential participants will be identified as possible study candidates with either chronic ETDD or baro-challenge ETDD, who have failed conservative management. At baseline, participants would undergo pure tone audiometry, tympanometry, and otoscopy. An ETDQ7, ad hoc work/activity impairment questionnaire, and EQ-5D-5L questionnaire would be completed. The patient's ability to equalize their middle ear pressure would be assessed by direct visualization of the tympanic membrane as the patient equalizes their middle ear pressure. For patients with baro-challenge ETDD, a baseline ad hoc questionnaire to quantify their symptoms will be completed as well.

Patients would then be randomized into BDET versus placebo groups. Patients in the experimental group undergoing BDET in-office will undergo dilation after anxiolytic pre-medication, nasal decongestion, as well as topical anesthesia of the lateral tympanic membrane, the eustachian tube orifice, and the nasal cavity. Patients randomized to the placebo group would undergo a similar procedure in-office, but without dilation of the eustachian tube. Patients in the experimental group with contraindication to in-office BDET will undergo BDET under general anesthetic in an operating room setting. The participants' first follow-up visit with the surgeon is at 6 weeks post-procedure, where patients in the placebo control group would be offered the option to cross-over into the BDET group. Follow up would also be repeated at 24 weeks and 52 weeks post-procedure.

ELIGIBILITY:
Inclusion Criteria (Chronic ETDD):

* >3 months of symptoms of ETDD (otalgia, ear pressure, muffled hearing, tinnitus, cracking or popping, feeling clogged) persistent at enrollment
* Persistence of symptoms despite >4 weeks INCS or >7d course of systemic steroid within 6 months from enrollment
* Documented Type B or C tympanogram at or within 6 months from enrollment
* ETDQ7 ≥ 2.1 at enrollment

Inclusion criteria (baro-challenge ETDD):

* >12 months of baro-challenge induced symptoms occurring at least every 4 months within the past year
* Symptoms include otalgia, ear pressure, muffled hearing, tinnitus, cracking or popping, feeling clogged, vertigo, or facial nerve palsy, which resolve within 3 days of pressure equalization.
* Failure of at least one of: topical/oral decongestant, pneumatization device, and/or pressure relief ear plugs.

Exclusion Criteria:

* Signs/symptoms of patulous eustachian tube dysfunction (autophony, tympanic membrane movement with breathing)
* Adjunctive surgical procedure needed (ex. septoplasty, tympanostomy tube)
* Presence of a tympanic membrane (TM) perforation or tympanostomy tube
* Fluctuating SNHL, AOM, grade IV TM retraction, or tympanosclerosis of >50% of the TM
* Uncontrolled sino-nasal disease, reflux, TMJ disorder, immunodeficiency, or allergies
* Known ICA dehiscence of the bony ET of the symptomatic ear
* Recent head and neck surgery within the past 3 months or planned procedure during study
* History of radiation to the head and neck
* History of craniofacial abnormality
* Prior ET intervention
* Psychiatric condition or cognitive impairment which precludes capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean Eustachian Tube Dysfunction Questionnaire (ETDQ7) score | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Score range 1-7, with higher score indicating more severe symptoms
Change in symptoms (ad hoc baro-challenge ETDD symptom questionnaire) | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Composite of quantitative and qualitative data points

SECONDARY OUTCOMES:
Change in tympanogram type and pressure at peak compliance | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Change from type C to A or type B to C or type B to A is considered improvement, and vice versa is considered deterioration. Pressure at peak compliance (continuous variable, where a value of zero is normal, and more negative values indicate worse ET function).
Change in audiogram (pure tone average thresholds) | 24 weeks
  Pure tone average thresholds measured at 500hz, 1khz, 2khz, and 4khz, where values below 25dB are normal, and higher values indicate worse hearing. Air-bone gap at 500hz, 1khz, 2khz, 4khz where normal value is 0dB, and higher values indicate worse conductive hearing.
Improvement in ability to equalize middle ear pressure | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Qualitative measure where inability to equalize middle ear pressures is a negative outcome.
Tympanic membrane position on otoscopy | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Qualitative measure where the tympanic membrane will be in a normal position, or in an abnormal retracted position.
Ad hoc work/activity impairment questionnaire score | 6 weeks, 24 weeks, and 52 weeks post-intervention
  Score range 1-7, with higher score indicating more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lui, MD, FRCSC, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Otology Clinic, Clinic 7A, South Health Campus, Calgary, Alberta
  - Sunnybrook Health Sciences Center, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No